CLINICAL TRIAL: NCT05189301
Title: The Differences in Oxygen Pulse Pattern During Maximum Incremental Exercise Test Between Norms and Patients With Chronic Obstructive Pulmonary Disease and With Chronic Heart Failure - the Possible Mechanisms
Brief Title: Oxygen Pulse and Its Curve Patterns in Male Patients With Heart Failure and Chronic Obstructive Pulmonary Disease With and in Healthy Men
Status: Completed | Type: Observational
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Ming-Lung Chuang, Visiting physician, Chung Shan Medical University
Other Study IDs: CSH-2019-C-030
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Outcome, Fatal
Keywords: exercise testing, oxygen pulse, chronic obstructive pulmonary disease, congestive heart failure, first pass study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CHF: CHF for chronic heart failure
  Interventions: Diagnostic Test: first pass study; Diagnostic Test: cardiopulmonary exercise testing
- COPD: COPD for chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: first pass study; Diagnostic Test: cardiopulmonary exercise testing
- control: control for normal controls
  Interventions: Diagnostic Test: first pass study; Diagnostic Test: cardiopulmonary exercise testing

INTERVENTIONS:
Diagnostic Test: first pass study — Radionuclide assessment of ventricular performance was performed (Symbia T2, Germany)
Diagnostic Test: cardiopulmonary exercise testing — to measured (mL/min, STPD), CO2 output ( ) (mL/min), and minute ventilation ( ) (L/min, BTPS) breath by-breath (MasterScreen CPX™, Germany)

SUMMARY:
Background: In non-invasive cardiopulmonary exercise testing (CPET), oxygen pulse (O2P) is defined as oxygen uptake divided by heart rate and is equal to the product of stroke volume and oxygen extraction by cells. As per, the O2P indicates the capability of oxygen consumption of whole body tissues and cells per heart beat. During exercise, the O2P changes can be deemed as the stroke volume changes as the oxygen extraction by muscle cells are normal. Hence, CPET-O2P can be non-invasively and continuously used to monitor the stroke volume changes during exercise. O2P value (i.e., % of predicted) is related to the severity and prognosis of heart failure and to the severity of constraint of the heart caused by exercise-induced hyperinflation or air trapping in patients with chronic obstructive pulmonary disease (COPD). However, O2P plateau pattern is not uncommonly encountered in the daily practice.

Hypothesis and aims: O2P patterns during incremental exercise are seldom investigated although they have been hypothesized that the plateau or decreasing patterns are related to myocardial failure or ischemia. In this proposal, the O2P patterns are to be thoroughly investigated: (1) the patterns in norms, patients with heart failure and COPD, (2) the relationship between the O2P pattern and cardiac function and/or myocardial ischemia in patients with heart failure and COPD. As yet there are no relative reports on the O2P pattern and its possible mechanisms in the literature, the results of the proposal might tremendously impact the interpretation strategy of CPET reports.

Methods: Multidisciplinary, prospective, comparative cross-sectional study is designed. Subjects aged from 40-85 years with the BMI of 18-28kg/m2 are to be enrolled: sample sizes of the norms, heart failure and COPD groups are 10, 20, and 20, respectively, equally distributed in two years. The definitions of COPD and heart failure with NYHA class I-III are according to the GOLD and ESC guidelines, respectively。All the three groups undergo CPET-NIRS, echocardiography, and the first pass and myocardial perfusion studies using Tc-99. The primary measurements are the O2P patterns and the cardiac function measured with echocardiography, the first pass and myocardial perfusion studies and air trapping in the lungs.。 Statistical analysis: For normal continuous data, t-test or ANOVA is used. For non-normal data, the Mann-Whitney test is used. The chi-square test or Fisher's exact test is used to compare the proportion of categorical variables between the two groups. A p value of less than .05 is considered to be statistically significant. Statistical procedures are performed using the SAS software package version 9.3.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 40-85 years with the BMI of 18-28kg/m2 are to be enrolled: sample sizes of the norms, heart failure and COPD groups are 10, 20, and 20, respectively, equally distributed in two years. All of the participants had been in a stable clinical condition for at least 1 month before participating in the study. None of the participants had contraindications for cardiopulmonary exercise tests (CPETs).

Exclusion Criteria:

* Participants with diabetes mellitus, uncontrolled hypertension, arrhythmia, cancer, liver, renal or autoimmune diseases, or anemia were excluded. However, participants with well controlled diabetes mellitus were included in the HFrEF/HFmrEF group as these conditions often co-exist. Physical activity was not encouraged or limited during the study period.

Age Groups: Child, Adult, Older Adult
Study Population: COPD. Participants with COPD were referred by pulmonologists, and they all had respiratory symptoms, risk factors and a post-bronchodilator forced expired volume in one second (FEV1)/forced vital capacity (FVC) of <0.7 in accordance with the Global Initiative for Chronic Lung Disease criteria.[23] Participants with a significant post-bronchodilator effect (increase in FEV1 >12% and 200 mL from baseline) were excluded.
  HFrEF/HFmrEF. Participants with HFrEF/HFmrEF who had reduced and mildly reduced EFs were referred by cardiologists, and they were enrolled if they had New York Heart Association functional class (NYHA) I-III, and risk factors. A left ventricular EF using two-dimensional echocardiography (2DLVEF) <45-50% was obtained within 2 months before or after commencing the study.[24] Normal controls. Healthy subjects were recruited among the hospital staff and the local community through personal contacts. They were free of known significant diseases.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
O2P and its patterns | one hour
  O2P value and its pattern were measured by exercise gas exchange.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Chuang, M.D., Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuang ML, Tsai CF, Ueng KC, Weng JH, Tsai MF, Lo CH, Chen GB, Sia SK, Chuang YT, Wu TC, Kao PF, Hsieh MJ. The Impact of Oxygen Pulse and Its Curve Patterns on Male Patients with Heart Failure, Chronic Obstructive Pulmonary Disease, and Healthy Controls-Ejection Fractions, Related Factors and Outcomes. J Pers Med. 2022 Apr 28;12(5):703. doi: 10.3390/jpm12050703. PMID 35629127